CLINICAL TRIAL: NCT00884377
Title: A Phase I/II Randomized Comparison of Localized Heat Therapy Versus Sodium Stibogluconate (Pentostam) for the Treatment of Old World Cutaneous Leishmaniasis (HSRRB Log No. A-12364)
Brief Title: Local Heat Therapy Versus Sodium Stibogluconate for the Treatment of Cutaneous Leishmaniasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Walter Reed Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-12364
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Results first posted 2017-07-14 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Cutaneous Leishmaniasis
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — Antimony Sodium Gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium stibogluconate intravenous (Active Comparator): 20 mg/kg/day Sodium stibogluconate intravenous
  Interventions: Drug: Sodium stibogluconate (Pentostam)
- ThermoMed device (Experimental): ThermoMed device, single heat treatment at 50 degrees Celsius
  Interventions: Device: ThermoMed

INTERVENTIONS:
Drug: Sodium stibogluconate (Pentostam) — intravenous 20 mg/kg/day for 10 days
  Other Names: Pentostam; WR 229,870
  Arms: Sodium stibogluconate intravenous
Device: ThermoMed — ThermoMed heat treatment device, one treatment
  Arms: ThermoMed device

SUMMARY:
This study serves to compare the effectiveness of treating cutaneous leishmaniasis with either intravenous sodium stibogluconate or direct heat therapy using the ThermoMed-TM device.

DETAILED DESCRIPTION:
A total of 56 Department of Defense health care beneficiaries, 18 years of age or older and diagnosed with cutaneous leishmaniasis, were planned to be treated with either intravenous sodium stibogluconate (Pentostam-TM) or the ThermoMed-TM device of Thermosurgery Technologies, Inc. at the Walter Reed Army Medical Center. Pentostam is the standard of care for this disease, but the i.v. administration and the many known side effects prompt the search for an improved method of treating this disease, especially for milder cases. This study compares the safety and efficacy of these two treatment approached.

ELIGIBILITY:
Inclusion Criteria:

* Department of Defense (DOD) Healthcare beneficiary
* Parasitologic diagnosis of cutaneous Leishmania infection

(Inclusion criteria for randomization includes that must be Leishmania major species)

* Willing to locate to WRAMC area during treatment and perform subsequent follow-up visits if needed

(If not active duty on orders, then the participant will bear the cost of food and lodging during the initial 10-day outpatient treatment period at Walter Reed Army Medical Center)

* Able to provide informed consent
* All participants (both male and female) must agree to take precautions not to become pregnant or father a child for at least 2 months after receiving sodium stibogluconate

Exclusion Criteria:

* Unable to provide informed consent
* Pregnancy (females of child bearing potential must have negative urine human chorionic gonadotropic hormone [HCG] within 48 hours of the start of infusion period)
* History of hypersensitivity to pentavalent antimonials
* Serious medical illness:

  1. QTc interval >/= 0.5 sec
  2. severe cardiac disease
  3. history of current pancreatitis
  4. liver failure or active hepatitis with transaminases >3X normal
  5. renal failure or creatinine >2.5
  6. thrombocytopenia (platelets <75,000)
  7. white blood cell count <2000
  8. hematocrit <25
  9. absence of palpable extremity pulses in the limb requiring treatment
* History of serious allergic reaction to local anesthetics
* Location of lesion not amenable to local therapy (such as close to eye, mucous membranes, face, cartilage)
* Presence of pacemaker and/or other implanted metallic devices
* Breast feeding
* Men unwilling to avoid fathering a child during and/or in the two months following receiving the treatment
* Women unwilling to avoid pregnancy for at least two months after receiving the treatment
* More than 20 lesions, or multiple lesions which in the opinion of the investigator would not be well treated with heat therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2004-02; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: COL Naomi Aronson, M.D., Principal Investigator — Uniformed Services University of the Health Sciences
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Aronson NE, Wortmann GW, Byrne WR, Howard RS, Bernstein WB, Marovich MA, Polhemus ME, Yoon IK, Hummer KA, Gasser RA Jr, Oster CN, Benson PM. A randomized controlled trial of local heat therapy versus intravenous sodium stibogluconate for the treatment of cutaneous Leishmania major infection. PLoS Negl Trop Dis. 2010 Mar 9;4(3):e628. doi: 10.1371/journal.pntd.0000628. PMID 20231896

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty Six subjects were recruited from the Infectious Disease Clinic at Walter Reed Army Medical Center from February 2004 to March 2009. At 2 months post-treatment, subjects assessed as having failed therapy were eligible for crossover to an alternate treatment.
Groups:
- Treatment With IV Sodium Stibogluconate: Subjects who had been randomized to the sodium stibogluconate group, received 10 days of treatment with sodium stibogluconate 20 mg/kg/day via intravenous infusions that were administered by health care personnel, generally in the WRAMC Infectious Disease Clinic or in the WRAMC infusion clinic.
- Treatment With Thermomed Device: Subjects randomized to the ThermoMed arm were given one treatment session using the ThermoMed device, Model 1.8, at 50°C. A heat treatment consisted of one or more 30-second heat applications of the ThermoMed device, with the number of applications dictated by lesion size. For lesions smaller than 2 mm, a treatment consisted of only one application of the ThermoMed device. For larger lesions, a treatment involved multiple overlapping applications of the device along an imaginary line that extended across the lesion and included approximately 4 mm of apparently healthy border skin. All of a subject's cutaneous leishmaniasis lesions, up to 20, were treated
Period: Overall Study
Arm/Group | Treatment With IV Sodium Stibogluconate | Treatment With Thermomed Device
Started | 28 (1 not treated because infecting parasite could not be confirmed as L. major on rapid PCR testing,) | 28 (1 was not treated due to concerns arising from the location of cutaneous leishmaniasis lesion)
Completed | 26 (1 received full course of therapy,withdrew consent before completion of the 12 month follow up) | 27
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Could not confirm diagnosis | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment With IV Sodium Stibogluconate | Treatment With Thermomed Device | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 28 | 56
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.0 (9.7) | 28.9 (8.3) | 27.9 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 27 | 28 | 55
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 60

OUTCOME MEASURES:

1. Primary Outcome: Equivalence of Efficacy Assessed by the Number of Participants With Clinical Cure
Description: Assess whether local heat therapy using the ThermoMed device was equivalent (clinical cure) in efficacy to 10 days of parenteral sodium stibogluconate. Clinical cure is defined as complete epithelialization of lesion. post-treatment, photographs of treated lesions were assessed for efficacy outcome by a consensus decision of leishmaniasis experts blinded as to each subject's study group. On the basis of these photo assessments, "clinical response" was assessed by lesion and by subject. In addition, an "overall response" was assigned ("healed" or "not healed") based on a combination of experts' photo assessments and subject interviews. Efficacy outcomes for the 2 study groups were compared using the Fishers exact test.
Time Frame: Assessment of cure is made at 2 months after treatment
Population: A sample size of 27 subjects per treatment group was planned based on the assumption that the cure rate in the heat treatment arm would be 73% (Navin et al., 1990), compared to a 99% cure rate in the sodium stibogluconate arm (Wortmann et al., 2002).
Measure: Count of Participants; unit: Participants
Groups:
- Sodium Stibogluconate: Sodium Stibogluconate group
- ThermoMed Device: ThermoMed device group
Arm/Group | Sodium Stibogluconate | ThermoMed Device
Number analyzed (Participants) | 28 | 28
Participants
  Healed | 22 | 18
  Not Healed | 5 | 9
  Not Applicable | 1 | 1
  Cured | 13 | 11
  Not Cured | 13 | 14
  Not Evaluable | 2 | 3

2. Secondary Outcome: Equivalence of Efficacy (Clinical Cure) of TheroMed Treatment vs Sodium Stibogluconate Assessed by the Number of Subjects With Clinical Cure
Description: Determine the equivalence of efficacy (clinical cure) of ThermoMed treatment vs sodium stibogluconate in clinical response of all skin lesions at 12 months. Clinical cure is defined as complete epithelialization of lesion. Post-treatment, photographs of treated lesions were assessed for efficacy outcome by a consensus decision of leishmaniasis experts blinded as to each subject's study group. On the basis of these photo assessments, "clinical response" was assessed by lesion and by subject. In addition, an "overall response" was assigned ("healed" or "not healed") based on a combination of experts' photo assessments and subject interviews. Efficacy outcomes for the 2 study groups were compared using the Fishers exact test.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Stibogluconate | ThermoMed Device
Number analyzed (Participants) | 28 | 28
Participants
  Healed | 25 | 23
  Not Healed | 2 | 4
  Not Applicable | 1 | 1
  Clincally Cured | 23 | 21
  Not Clinically Cured | 2 | 2
  Not Evaluable | 3 | 5

3. Secondary Outcome: Number of Participants With Solicited Adverse Events
Description: To compare the toxicity profiles of ThermoMed treatment versus parenteral sodium stibogluconate therapy thru specific solicited adverse events
Time Frame: Days 3, 7 and 10
Population: Data ia showing only subjects with specified solicited symptoms on Days 3, 7 and 10. Collective count of participants for SSG is 53 and 28 for ThermoMed over all reported days.
Measure: Number; unit: subjects showing specified symptoms
Groups:
- Sodium Stibogluconate: Sodium Stibogluconate Groups
- ThermoMed Treatment: ThermoMed Treatment Groups
Arm/Group | Sodium Stibogluconate | ThermoMed Treatment
Number analyzed (Participants) | 28 | 28
subjects showing specified symptoms
  Myalgias : Day 3 | 4 | 1
  Myalgias : Day 7 | 3 | 0
  Myalgias : Day 10 | 5 | 0
  Arthralgias : Day 3 | 4 | 2
  Arthralgias : Day 7 | 11 | 2
  Arthralgias : Day 10 | 7 | 2
  Nausea : Day 3 | 3 | 1
  Nausea : Day 7 | 4 | 0
  Nausea : Day 10 | 1 | 1
  Vomiting : Day 3 | 1 | 0
  Vomiting : Day 7 | 2 | 0
  Vomiting : Day 10 | 0 | 0
  Abdominal Pain : Day 3 | 2 | 0
  Abdominal Pain : Day 7 | 3 | 0
  Abdominal Pain : Day 10 | 2 | 1
  Headache : Day 3 | 7 | 2
  Headache : Day 7 | 9 | 2
  Headache : Day 10 | 5 | 2
  Diarrhea : Day 3 | 2 | 1
  Diarrhea : Day 7 | 3 | 0
  Diarrhea : Day 10 | 3 | 1
  Rash : Day 3 | 2 | 1
  Rash : Day 7 | 2 | 0
  Rash : Day 10 | 3 | 1
  Fever : Day 3 | 0 | 0
  Fever : Day 7 | 2 | 0
  Fever : Day 10 | 0 | 0
  Fatigue : Day 3 | 17 | 3
  Fatigue : Day 7 | 11 | 1
  Fatigue : Day 10 | 9 | 3
  Chest Pain : Day 3 | 1 | 0
  Chest Pain : Day 7 | 0 | 0
  Chest Pain : Day 10 | 0 | 0
  Other : Day 3 | 3 | 2
  Other : Day 7 | 6 | 5
  Other : Day 10 | 2 | 7

4. Secondary Outcome: Immune Response, Based on T-Cell Population Before Treatment, and Day 10 Following Treatments
Description: Evaluate the immune response (T-Cell population) to Leishmania before treatment, and at 10 days, in recipients of localized heat therapy vs systemic sodium stibogluconate. Days 1 and 10 are presented in columns.
Time Frame: day 1 and day 10
Population: Populations of T-cells CD3+CD8, CD19, CD16+CD56 on study days 1 and 10
Measure: Mean (95% Confidence Interval); unit: populations of T-cells
Groups:
- Study Day 1: Sodium Stibogluconate: Day 1: Sodium Stibogluconate group
- Study Day 10: Sodium Stibogluconate: Day 10: Sodium Stibogluconate group
- Study Day 1: ThermoMed: Day 1: TherrmoMed group
- Study Day 10: ThermoMed: Day 10: ThermoMed group
Arm/Group | Study Day 1: Sodium Stibogluconate | Study Day 10: Sodium Stibogluconate | Study Day 1: ThermoMed | Study Day 10: ThermoMed
Number analyzed (Participants) | 27 | 26 | 27 | 27
populations of T-cells
  ABS CD3+CD8 (cells/uL) | 515.89 [97.00 to 950.00] | 534.19 [228.00 to 1150.00] | 368.74 [63.00 to 1092.00] | 500.15 [259.00 to 754.00]
  ABS CD19 (cells/uL) | 375.37 [121.00 to 806.00] | 328.27 [145.00 to 613.00] | 213.85 [76.00 to 447.00] | 274.70 [172.00 to 513.00]
  ABS CD16+CD56 (cells/uL) | 196.52 [66.00 to 474.00] | 207.62 [111.00 to 406.00] | 137.74 [49.00 to 603.00] | 221.96 [122.00 to 482.00]

5. Secondary Outcome: Immune Response, Based on Percent of T-Cell Population Before Treatment, and Day 10 Following Treatments
Description: as for outcome 4
Time Frame: day 1 and day 10
Population: Percent of T-cells CD3+CD8, CD19, CD16+CD56 on study days 1 and 10
Measure: Mean (95% Confidence Interval); unit: % of T-cells
Arm/Group | Study Day 1: Sodium Stibogluconate | Study Day 10: Sodium Stibogluconate | Study Day 1: ThermoMed | Study Day 10: ThermoMed
Number analyzed (Participants) | 27 | 26 | 27 | 27
% of T-cells
  CD3+CD8 (%) | 25.07 [9.00 to 41.00] | 26.54 [16.00 to 38.00] | 25.67 [10.00 to 40.00] | 26.85 [15.00 to 38.00]
  CD19 (%) | 17.96 [8.00 to 37.00] | 16.73 [8.00 to 31.00] | 15.30 [8.00 to 32.00] | 15.11 [9.00 to 25.00]
  CD16+CD56 (%) | 9.67 [4.00 to 16.00] | 10.73 [6.00 to 19.00] | 9.81 [3.00 to 24.00] | 11.74 [6.00 to 25.00]

6. Secondary Outcome: Feasibility of a L. Major Species Specific Polymerase Chain Reaction as a Rapid Diagnostic Device in the Context of a Treatment Trial
Description: Evaluate the feasibility of using species-specific PCR as a rapid diagnostic assay for L. major infection. The comparator modalities were: histopathology (identification of amastigotes); speciation determined through culture and isoenzyme analysis; and genus and species-specific PCR. Species PCR testing was performed at baseline to allow for the identification of L. major as each subject's infecting parasite. If an L. major infection could not be confirmed in a subject's lesion(s), then that subject could not be treated under this protocol.
Time Frame: at baseline before treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Stibogluconate | ThermoMed Device
Number analyzed (Participants) | 28 | 28
Participants
  Histopathology: Amastigotes absent | 10 | 6
  Histopathology: Amastigotes present | 18 | 22
  Culture: Not done | 4 | 5
  Culture: Unknown | 0 | 1
  Culture: Negative | 6 | 4
  Culture: Positive | 18 | 18
  Culture/Isoenzyme Analysis: L.major = Positive | 12 | 12
  Culture/Isoenzyme analysis: Unknown Leish species | 2 | 3
  Culture/Isoenzyme analysis: Not done | 4 | 4
  PCR (Genus) = Positive for Leish genus | 28 | 28
  PCR (Species) = Positive for L.major species | 27 | 28
  PCR (Species) = Unknown | 1 | 0

ADVERSE EVENTS:
Time Frame: Day 1-10 AEs were documented daily. After day 10, AE surveillance was performed via subject interviews at 2, 6 and 12 months (window of 10-24 months) post-treatment.
Arm/Group | Sodium Stibogluconate Intravenous | ThermoMed Device
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 5/28 | 2/28
Other Adverse Events (participants affected / at risk) | 28/28 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Stibogluconate Intravenous (N=28) | ThermoMed Device (N=28)
Accute gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Severe; resolved; unrelated
Osteoarthritis, left acromioclavicular joint (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Moderate; resolved; unrelated
Injury, spine trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Severe; resolved; unrelated
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0) — Moderate; resolved; unrelated
Transanal resection of carcinoid tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Moderate; resolved; unrelated
Crohn's disease exacerbation (Immune system disorders) | 0 (0) | 1 (1) — Moderate; resolved; unrelated
Basal cell carcinoma, superficial (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Mild; resolved; unrelated
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Stibogluconate Intravenous (N=28) | ThermoMed Device (N=28)
Lesion site blister (Skin and subcutaneous tissue disorders) | 0 (0) | 25 (25) — Local (lesion related)
No blanching with pressure (Vascular disorders) | 1 (1) | 18 (18) — Local (lesion related)
Site erythema (Skin and subcutaneous tissue disorders) | 5 (5) | 21 (21) — Local (lesion related)
Site eschar (Injury, poisoning and procedural complications) | 9 (9) | 25 (25) — Local (lesion related)
Site infection (Infections and infestations) | 1 (1) | 5 (5) — Local (lesion related)
Site keloid formation (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) — Local (lesion related)
Site pain (General disorders) | 2 (2) | 11 (11) — Local (lesion related)
Site papules (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3) — Local (lesion related)
Site plaque (Injury, poisoning and procedural complications) | 10 (10) | 7 (7) — Local (lesion related)
Site pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (6) — Local (lesion related)
Satellite lesions (Infections and infestations) | 2 (2) | 3 (3) — Local (lesion related)
Site scaley (Skin and subcutaneous tissue disorders) | 11 (11) | 6 (6) — Local (lesion related)
Site tenderness (General disorders) | 2 (2) | 5 (5) — Local (lesion related)
Site ulcer (Injury, poisoning and procedural complications) | 11 (11) | 14 (14) — Local (lesion related)
Site verrucous (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) — Local (lesion related)
Site weeping (General disorders) | 2 (2) | 23 (23) — Local (lesion related)
Site oedema (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) — Local (lesion related)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) — General (non-lesion related)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 (3) | 4 (4) — General (non-lesion related)
Tachycardia (Cardiac disorders) | 5 (5) | 3 (3) — General (non-lesion related)
Ventricular hypertrophy (Cardiac disorders) | 3 (3) | 0 (0) — General (non-lesion related)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 1 (1) — General (non-lesion related)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 2 (2) — General (non-lesion related)
Nausea (Gastrointestinal disorders) | 8 (8) | 2 (2) — General (non-lesion related)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) — General (non-lesion related)
Chest pain (General disorders) | 3 (3) | 0 (0) — General (non-lesion related)
Fatigue (General disorders) | 28 (28) | 7 (7) — General (non-lesion related)
Pyrexia (General disorders) | 4 (4) | 0 (0) — General (non-lesion related)
Site extravasation (General disorders) | 5 (5) | 0 (0) — General (non-lesion related)
Chemical hepatitis (Hepatobiliary disorders) | 3 (3) | 0 (0) — General (non-lesion related)
Amylase increased (Investigations) | 19 (19) | 0 (0) — General (non-lesion related)
Lipase increased (Investigations) | 23 (23) | 0 (0) — General (non-lesion related)
ALT increased (Investigations) | 13 (13) | 0 (0) — General (non-lesion related)
AST increased (Investigations) | 9 (9) | 0 (0) — General (non-lesion related)
EKG T-wave abnormal (Investigations) | 2 (2) | 3 (3) — General (non-lesion related)
QRS axis abnormal (Investigations) | 4 (4) | 4 (4) — General (non-lesion related)
WBC decreased (Investigations) | 9 (9) | 2 (2) — General (non-lesion related)
Eosinophil count increased (Investigations) | 2 (2) | 3 (3) — General (non-lesion related)
Monocyte count increased (Investigations) | 7 (7) | 1 (1) — General (non-lesion related)
Platelet count decreased (Investigations) | 8 (8) | 2 (2) — General (non-lesion related)
Albumin decreased (Investigations) | 6 (6) | 3 (3) — General (non-lesion related)
Chloride increased (Investigations) | 5 (5) | 1 (1) — General (non-lesion related)
Creatine phosphokinase increased (Investigations) | 2 (2) | 3 (3) — General (non-lesion related)
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 (22) | 6 (6) — General (non-lesion related)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) — General (non-lesion related)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (12) | 1 (1) — General (non-lesion related)
Headache (Nervous system disorders) | 21 (21) | 6 (6) — General (non-lesion related)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) — General (non-lesion related)
Rash (Skin and subcutaneous tissue disorders) | 7 (7) | 2 (2) — General (non-lesion related)
Dizziness (Vascular disorders) | 3 (3) | 1 (1) — General (non-lesion related)
Fever (General disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No